CLINICAL TRIAL: NCT01784406
Title: Person-centred Support for Women in the Follow-up Period After Surgical Treatment for Gynaecological Cancer - a Randomised Controlled Trial
Brief Title: Person-centred Support for Women After Treatment for Gynaecological Cancer
Acronym: PESU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mette Linnet Olesen, Ph.d student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-4-2012-FSP(94)
Record Dates: First submitted 2013-02-03; First posted 2013-02-05 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Malignant Female Reproductive System Neoplasm; Follow-up; Supportive Care; Psychosocial Circumstances; Survivorship
Keywords: Self-management intervention; Psychosocial care; Autonomy-supportive; Gynaecological cancer survivors; Guided self-Determination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autonomy-supportive counselling (Experimental): 2-4 autonomy-supportive conversations with an experienced nurse, educated both theoretically and practically in the method Guided Self-Determination that includes specific "reflection sheets" and use of advanced communication; in addition to standard care.
  Interventions: Behavioral: Autonomy supportive counselling
- Control (No Intervention): Standard of care.

INTERVENTIONS:
Behavioral: Autonomy supportive counselling
  Arms: Autonomy-supportive counselling

SUMMARY:
Women treated for gynaecological cancer perceive many difficulties in life on the personal, social, and physical levels. Today they are offered a 3 to 5 year follow-up programme at the hospital where the main purpose is to improve survival. However, the women are very nervous before follow-up visits and although they feel safe about them, they express that their needs of psychosocial care and self-management support are not fulfilled.

The proposed study will test a person-centred intervention tailored the women's needs in a randomised controlled trial. The intervention will be based on the method Guided Self Determination (GSD), which has proved able to realize empowerment in practice in relationships between patients and healthcare professionals. GSD involves systematic use of condition-adjusted worksheets ('reflection sheets'), and advanced professional communication. Using reflection sheets filled out by each woman as the starting point for communication, problem solving will be tailored her personal needs. We expect that the intervention has the potential to support the women in better managing specific complications and difficulties related to concerns about recovery, body perception, fertility and establishment of intimate relations with their partner, all aspects important for the women's quality of life in the follow-up period after cancer diagnosis and treatment. The study will be the first to test GSD in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Women only surgically treated for cervix, ovarian (including borderline tumors), endometrial or vulva cancer, who attend follow up at the Gynaecological Department at The University Hospital Rigshospitalet in Copenhagen.
* The women should read, write and understand the danish language.

Exclusion criteria:

* Known recurrence.
* Participation in the preliminary pilotstudy.
* Health related problems both physical or psychological, that prevent participation. For example cognitive impairment, or patients with psychiatric diseases that is estimated to require nurses with competences within the psychiatric speciality.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Primary Outcome: Quality of life measured by the scale Quality of life- Cancer Survivors (QOL-CS) | 9 months after randomisation
  +/- one week for practical reasons

SECONDARY OUTCOMES:
Quality of Life measured by the scale Quality of Life Cancer Survivors- (QOL-CS) | 3 months after randomisation
  +/- one week for practical reasons
Changes in Quality of life in the two groups | 9 months
  Quality of life at 9 months minus the quality of life at the time of randomisation.
Positive and negative impact of cancer measured by Impact of Cancer version 2 (IOCv2) | 3 and 9 months after randomisation
  +/- one week for practical reasons
Self-esteem measured by Rosenbergs Self Esteem Scale | 3 and 9 months after randomisation
  +/- one week for practical reasons
Anxiety and depression measured by Hospital Anxiety and Depression Scale (HADS) | 3 and 9 months from randomisation
  Also used as screening instrument baseline.
  +/- one week for practical reasons
Autonomy-supportive relationship between patient and health care professionals measured by Health Care Climate Questionnaire (HCCQ) | 3 and 9 months from randomisation
  +/- one week for practical reasons
Distress measured by Distress Thermometer(DT). | 3 and 9 months from randomisation
  Also used as screening instrument baseline.
  +/- one week for practical reasons.
Symptom monitoring and recognition | 3 and 9 months after randomisation (+/- one week for practical reasons)
  Womens ability to know what symptoms to monitor and react to in case of recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Gynaecological Department, Juliane Marie Centret,Copenhagen University Hospital Rigshospitalet, Copenhagen, Copenhagen Ø, Denmark

REFERENCES:
- See also: Statistical analysis plan — http://www.rigshospitalet.dk/NR/rdonlyres/37378D7E-6E5E-4BC7-B46A-1969CB0DEE8D/0/June2014StatisticalanalysisplanPersoncenteredsupportforwomenaftertreatmentforgynaecologicalcancer.pdf
- See also: Copenhagen University Hospital, Rigshospitalet has changed to a new web system therefore a new url adress/Statistical analysis plan — http://www.rigshospitalet.dk/afdelinger-og-klinikker/julianemarie/forskningsenheden-kvinders-og-boerns-sundhed/forskning/forskningsprojekter-i-enheden/Documents/June2014StatisticalanalysisplanPersoncenteredsupportforwomenaftertreatmentforgynaecologicalcancer.pdf